CLINICAL TRIAL: NCT03116425
Title: Personalized Non-invasive Neuromodulation by rTMS for Chronic and Treatment Resistant Catatonia - A Proof of Concept Study
Brief Title: Personalized Non-invasive Neuromodulation by rTMS for Chronic and Treatment Resistant Catatonia
Acronym: RETONIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 6441
Record Dates: First submitted 2017-03-22; First posted 2017-04-17 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Schizophreniform Catatonia; Treatment Resistant
Keywords: Precision Medicine; Functional Neuroimaging; Transcranial Magnetic Stimulation, Repetitive; Transcranial Direct Current Stimulation; Monocentric; Comparative balanced, randomized; double-blind cross-over 3 Arms Study
MeSH Terms: conditions — Catatonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum 1 - Premotor (Experimental): The target region will be defined by comparing the rCBF scan of the patient to a control population (n = 38). rCBF will be measured using the QUIPS2 arterial spin labeling sequence on a Siemens 3T Verio.
  The network including the premotor region will be targeted. The therapeutic protocol will be design to correct the rCBF anomaly.
  Interventions: Device: Individualized rTMS on VERUM 1's region or network; Procedure: Individualized rTMS on VERUM 1's region or network
- Verum 2 - Prefrontal (Experimental): The target region will be defined by comparing the rCBF scan of the patient to a control population (n = 38). rCBF will be measured using the QUIPS2 arterial spin labeling sequence on a Siemens 3T Verio.
  The network including the prefrontal region will be targeted. The therapeutic protocol will be design to correct the rCBF anomaly.
  Interventions: Device: Individualized rTMS on VERUM 2's region or network; Procedure: Individualized rTMS on VERUM 2's region or network
- Placebo (Active Comparator): Stimulation of a region with normal rCBF and putatively unrelated to catatonic symptoms (parietal cortex).
  Interventions: Device: Individualized rTMS on PLACEBO region; Procedure: Individualized rTMS on PLACEBO region

INTERVENTIONS:
Device: Individualized rTMS on VERUM 1's region or network — To increase cortical rCBF, iTB (intermittent theta burst) will be used: triplet at 50 Hz repeated at 5 Hz in trains of 2 sec with an inter-train interval of 8 sec.
  To decrease cortical rCBF, cTB (continuous theta burst) will be used: triplet at 50 Hz repeated at 5 Hz in trains of 40 sec. Intensity 120% of passive threshold (or 150% of active threshold).
  Stimulation protocol will be used up to 5 times per session to allow a reasonable regional or network coverage.
  Patients will have 4 sessions per day on 5 successive days per arm.
  Other Names: Putative premotor region or network
  Arms: Verum 1 - Premotor
Device: Individualized rTMS on VERUM 2's region or network — To increase cortical rCBF, iTB (intermittent theta burst) will be used: triplet at 50 Hz repeated at 5 Hz in trains of 2 sec with an inter-train interval of 8 sec.
  To decrease cortical rCBF, cTB (continuous theta burst) will be used: triplet at 50 Hz repeated at 5 Hz in trains of 40 sec. Intensity 120% of passive threshold (or 150% of active threshold).
  Stimulation protocol will be used up to 5 times per session to allow a reasonable regional or network coverage.
  Patients will have 4 sessions per day on 5 successive days per arm.
  Other Names: Putative prefrontal region or network
  Arms: Verum 2 - Prefrontal
Device: Individualized rTMS on PLACEBO region — Region will be modulated up or down according to the stimulation protocol used in VERUM 1 and 2 conditions.
  Stimulation will be replicated up to 5 times per session. Patients will have 4 sessions per day on 5 successive days per arm.
  Other Names: (One per line)
  Arms: Placebo
Procedure: Individualized rTMS on VERUM 1's region or network — To increase cortical rCBF, iTB (intermittent theta burst) will be used: triplet at 50 Hz repeated at 5 Hz in trains of 2 sec with an inter-train interval of 8 sec.
  To decrease cortical rCBF, cTB (continuous theta burst) will be used: triplet at 50 Hz repeated at 5 Hz in trains of 40 sec. Intensity 120% of passive threshold (or 150% of active threshold).
  Stimulation protocol will be used up to 5 times per session to allow a reasonable regional or network coverage.
  Patients will have 4 sessions per day on 5 successive days per arm.
  Other Names: Putative premotor region or network
  Arms: Verum 1 - Premotor
Procedure: Individualized rTMS on VERUM 2's region or network — To increase cortical rCBF, iTB (intermittent theta burst) will be used: triplet at 50 Hz repeated at 5 Hz in trains of 2 sec with an inter-train interval of 8 sec.
  To decrease cortical rCBF, cTB (continuous theta burst) will be used: triplet at 50 Hz repeated at 5 Hz in trains of 40 sec. Intensity 120% of passive threshold (or 150% of active threshold).
  Stimulation protocol will be used up to 5 times per session to allow a reasonable regional or network coverage.
  Patients will have 4 sessions per day on 5 successive days per arm.
  Other Names: Putative prefrontal region or network
  Arms: Verum 2 - Prefrontal
Procedure: Individualized rTMS on PLACEBO region — Region will be modulated up or down according to the stimulation protocol used in VERUM 1 and 2 conditions.
  Stimulation will be replicated up to 5 times per session. Patients will have 4 sessions per day on 5 successive days per arm.
  Arms: Placebo

SUMMARY:
Investigators hypothesize that personalizing rTMS targets using functional MRI will allow to improve symptoms of patients suffering from chronic catatonia.

DETAILED DESCRIPTION:
Two dysfunctional networks or regions will be chosen (verum 1 and 2) based on their abnormal rCBF. In line with the symptoms, dorso-lateral prefrontal and premotor regions are expected to be chiefly concerned. A normal region regarding its rCBF will be used as placebo. Targets will be stimulated using intermittent or continuous theta-burst according to the rCBF anomaly as an attempt to "normalize" their activity. The coil will be positioned using a robotic device under the control of a neuronavigation system in order to deliver a homogeneous stimulation. Using a balanced blinded randomized cross-over design, patients will be stimulated on 5 consecutive days (4 sessions per day) and evaluated pre-, post-stimulation and 1 month after. In this pilot study the primary outcome measures will be the clinical global impression scale whereas MRI will insure that stimulations achieved the correction of the rCBF anomalies. Secondary outcome measures will include personalized target symptom scales, and scales for catatonic, apathic and obsessive-compulsive symptoms.

ELIGIBILITY:
Inclusion criteria:

* Aged from 18 to 70 Y
* Affiliated to the health insurance
* Having signed an informed consent
* Suffering from catatonia according to the DSM5, unremitted since > 2Y
* Unresponsive or incomplete remission after at least one trial of benzodiazepine and/or Electroconvulsivotherapy
* Treatment stable for > 6 weeks

Exclusion criteria:

* Contraindication for MRI, rTMS or tDCS: non-removable ferromagnetic body, prosthesis, pacemaker, medication delivered by an implanted pump clip or vascular stent, heart valve or ventricular shunt, seizure disorders, skin pathology in the region of tDCS electrode placement.
* Pregnancy
* Severe and non-stabilized somatic pathology
* Patients deprived of liberty or hospitalized without their consent
* Patients unable to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Clinical global impression (change in severity and improvement) | In term of percentage reduction in symptoms, difference between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention

SECONDARY OUTCOMES:
Change in personalized daily visual analogical scales assessing the core symptoms. | Points results will be averaged over the 4 days before and after each therapeutic arm.
  This scale has been validated
Change in Bush and Francis Catatonia Rating Scale. | Points involvement in scale between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  This scale has been validated.
Change in psychosis: PANSS. | Points involvement in scale between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  This scale has been validated.
Change in depression: Calgary Depression Scale. | Points involvement in scale between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  This scale has been validated.
Change in apathy: actimetry, apathy inventory and apathy evaluation scale. | Points involvement in scale between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  This scale has been validated.
Change in obsessive compulsive symptoms: Brief Obsessive Compulsive Scale | Points involvement in scale between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  This scale has been validated.
Change in obsessive compulsive symptoms: Cambridge-Exeter Repetitive Thought Scale. | Points involvement in scale between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  This scale has been validated.
Change in quality of life for the patient (SF36) | Points involvement in scale between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  All these scales have been validated.
Change in the helping person ("Zarit scale") | Points involvement in scale between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  This scale has been validated.
Change in functioning: Global Assessment of Functioning (GAF scale) | Points involvement in scale between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  This scale has been validated.
Change in functioning: WHODAS 2.0. | Points involvement in scale between before (assessed on D1) and after (assessed on D5 to 7) and at 1 month after each therapeutic protocol (D = day of the beginning of the protocol)
  This scale has been validated.

OTHER OUTCOMES:
Change of rCBF anomalies | Points involvement in scale between before (assessed once between D-7 to -1) and after (assessed once between D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol).
  The target region will be defined by comparing the rCBF scan of the patient to a control population (n = 38). rCBF will be measured using the average of 2 ∙ 3 (=6) measures of rCBF using QUIPS2 arterial spin labeling sequence on a Siemens 3T Verio. We will compare the rCBF change of the target region before and after the therapeutic protocol between the different procedures (ANOVA).

CONTACTS AND LOCATIONS:
Overall Officials: Jack FOUCHER, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- CEMNIS, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No